CLINICAL TRIAL: NCT07372157
Title: Investigation of the Effectiveness of Neuromuscular Control-Based Exercises Combined With Aerobic and Strength Training Exercises on Balance in Overweight and Obese Individuals
Brief Title: Neuromuscular Balance Exercise Effects in Overweight and Obese Individuals
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, M. Gulden Polat, Professor of Physiotherapy and Rehabilitation, Marmara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 130.2024fbu
Record Dates: First submitted 2025-12-18; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-12

CONDITIONS: Overweight and Obesity
Keywords: Obesity; Exercise; Neuromuscular control; Quality of life; Postural stability
MeSH Terms: conditions — Overweight; Obesity; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to either a control group or an intervention group, and both groups are followed in parallel throughout the study period.
Masking Description: This is an open-label study with no blinding of participants or investigators.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Participants in the control group are individuals with obesity or overweight who receive a standardized exercise program that includes aerobic and strength training exercises. The program is performed three times per week over an eight-week period.
  Interventions: Behavioral: Aerobic and strength training
- Intervention group (Experimental): Participants in the intervention group consist of individuals with obesity or overweight who receive the same aerobic and strength training program as the control group, with the addition of neuromuscular balance exercises. The intervention is performed three times per week for eight weeks.
  Interventions: Behavioral: Aerobic and strength training; Behavioral: Neuromuscular balance exercises

INTERVENTIONS:
Behavioral: Aerobic and strength training — The aerobic and strength training program consists of supervised exercise sessions performed three days per week for eight weeks. Aerobic exercises are conducted at a moderate intensity, and strength training targets major muscle groups using body weight and resistance-based exercises. Each session is structured to include warm-up, main exercise components, and cool-down phases.
Behavioral: Neuromuscular balance exercises — Neuromuscular balance exercises are added to the standard exercise program and are designed to improve postural control and balance. The exercises include progressive static and dynamic balance tasks and are performed three times per week for eight weeks under supervision.
  Arms: Intervention group

SUMMARY:
This randomized controlled study aims to evaluate the effects of adding neuromuscular balance exercises to exercise programs on functional capacity, balance, and physical fitness in individuals with obesity. Forty participants will be randomly assigned to either a control group receiving aerobic and strength training exercises or an intervention group receiving aerobic and strength training combined with neuromuscular balance exercises. Both exercise programs will be conducted three times per week for eight weeks. Functional capacity, balance, and physical fitness outcomes will be assessed at baseline and after the intervention period. The findings are expected to contribute to the integration of balance-focused exercises into rehabilitation programs for individuals with obesity.

DETAILED DESCRIPTION:
This project will begin with initial assessments of volunteers to examine the effects of balance exercises on postural control and neuromuscular connections in obesity treatment. A multimodal exercise program (neuromuscular balance exercises, aerobic training, and resistance training) will be designed for individuals with obesity, and its effects on physical function, balance impairment, and weight management will be evaluated. In the first phase, participants' static and dynamic balance will be analyzed using clinical scales. In the second phase, an 8-week multimodal exercise program will be implemented, and the outcomes will be comparatively examined in relation to the weight loss process.

The study aims to provide scientific data to support the individualization of exercise programs by examining postural balance adaptations in response to changes in body composition during weight loss. The findings are expected to contribute to more comprehensive physical activity approaches in obesity management and to guide clinical applications.

This study adds a different perspective by evaluating the functional benefits of neuromuscular-based balance exercises in addition to traditional aerobic and strength training exercises. The assessment, conducted in individuals with obesity who have experienced weight loss, is expected to provide important findings for the interpretation and discussion of outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Having a BMI of 25-35 kg/m2
* Not having undergone any surgical operation in the last 6 months

Exclusion Criteria:

* Any musculoskeletal disorder or systemic disease that would prevent exercise
* Balance problems due to any disease that could prevent exercise
* Psychiatric or neurological disease affecting cooperation and cognitive functions
* Acute pain for any reason
* Chest pain
* History of myocardial infarction within the last year
* Congestive heart failure
* Patient's inability to adhere to treatment

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-15 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Dynamic Balance Performance (Four Step Square Test) | Baseline, at the 4th weeks and at the end of 8 weeks
  Dynamic balance will be assessed using the Four Step Square Test, which measures the time (in seconds) required to complete a multidirectional stepping sequence.
Postural Control (Functional Reach Test) | Baseline, Week 4, and Week 8
  Postural control will be evaluated using the Functional Reach Test, which measures the maximal forward reach distance (in centimeters) while maintaining a fixed base of support.
Walking Endurance (2-Minute Walk Test) | Baseline, at the 4th weeks and at the end of 8 weeks
  Walking endurance will be assessed using the 2-Minute Walk Test, which measures the total distance walked in meters over a two-minute period.
Lower Extremity Functional Strength (30-Second Chair Stand Test) | Baseline, Week 4, and Week 8
  Lower extremity functional strength will be evaluated using the 30-Second Chair Stand Test, which measures the number of full stands completed within 30 seconds.

SECONDARY OUTCOMES:
Health-Related Quality of Life Assessed by the Short Form-12 (SF-12) | Baseline, at the 4th weeks and at the end of 8 weeks
  Health-related quality of life will be evaluated using the Short Form-12 (SF-12) Health Survey, which assesses physical and mental health components.

CONTACTS AND LOCATIONS:
Overall Officials: Mine Gülden G Polat, PhD, Principal Investigator — Marmara University Faculty of Health Sciences
Locations (1):
- Fatih Sultan Mehmet Training and Research Hospital, Diabetes and Obesity Treatment Center, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.